CLINICAL TRIAL: NCT05254886
Title: Identification and Management of Comorbidities and Extra-intestinal Manifestations in Crohn's Disease: the NEMO Nurse-led Program
Acronym: NEMO-Nurse
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr Laurent PEYRIN-BIROULET, Principal Investigator, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021PI157
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine practice (No Intervention): Patients who benefit from the classic management of CD (i.e. clinical + biological ± radiological ± endoscopic follow-up ± therapeutic education program).
- Routine practice + nurse-led program (Experimental): Patients who receive, in addition to routine practice, a single nursing consultation dedicated to the identification and management of comorbidities and EIMs in CD at the inclusion visit.
  Interventions: Other: NEMO nurse-led program

INTERVENTIONS:
Other: NEMO nurse-led program — The NEMO nurse-led program will consist of a single nursing consultation conducted on the day of the inclusion visit during which the nurse will:
  * Report the presence of pre-existing comorbidities/EIMs
  * Detect the presence of risk factors
  * Implement recommendations for the detection and/or management of comorbidities/EIMs.
  Arms: Routine practice + nurse-led program

SUMMARY:
Crohn's disease (CD) is a chronic inflammatory disease of the gastrointestinal (GI) tract. Although inflammation is predominantly expressed in the GI tract, extra-intestinal manifestations (EIMs) are so frequent that the concept of systemic disease is now widely accepted. Moreover, similar to other chronic diseases, patients with CD can be affected by other unrelated diseases which are called comorbidities.

Although no specific guidelines on comorbidity and EIMs in CD are available, data from other immune-mediated diseases support the use of nurse-led programs to improve the cost-effectiveness for the management of cardiovascular risk factors, increase rates of pneumococcal vaccination in high-risk patients, provide preventive measures against osteoporosis and increased fracture risk in older women.

The investigators believe that such an initiative can be conducted for CD patients by developing a CD-specific nurse-led program. Moreover, it has been shown that CD patients highly appreciate the "communicator role" and "skilled companionship" performed by nurses to fulfill their needs for attention to the "complete picture".

Therefore, the investigators hypothesize that a nurse-led program would increase the number of measures taken to treat or identify EIMs and/or comorbidities in CD patients and thus revolutionize their management.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of CD with a minimum disease duration of 3 months
* CD considered by the treating gastroenterologist to have been stable for at least 3 months
* No surgery planned within 6 months after the inclusion visit

Exclusion Criteria:

* Subject unable to attend all the study visits or comply with study procedures.
* Subject unwilling or not able to understand or sign the informed consent.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 198 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of measures taken by a physician in order to prevent or treat comorbidities and EIMs associated with CD | 6 months
Number of measures taken by a physician in order to prevent or treat comorbidities and EIMs associated with CD | 18 months

SECONDARY OUTCOMES:
Number of measures taken by a physician for each comorbidity and EIM associated with CD in order to prevent or treat them | 6 months
Number of measures taken by a physician for each comorbidity and EIM associated with CD in order to prevent or treat them | 18 months
Percentage of patients who comply with recommendations issued by the nurse following completion of the NEMO nurse-led program | 6 months
Percentage of patients who comply with recommendations issued by the nurse following completion of the NEMO nurse-led program | 18 months
Level of patient satisfaction with the NEMO nurse-led program | 6 months
  Assessment with a Satisfaction Questionnaire. Answer options are presented on a 4-item Likert scale and ranges from 1 ('Not at all satisfied') to 4 ('Very satisfied'). Total score is summed up and ranges from 14 to 56, higher score indicating higher levels of satisfaction.
Frequency of comorbidities and EIMs, confirmed by a medical specialist, associated with CD | 6 months
Frequency of comorbidities and EIMs, confirmed by a medical specialist, associated with CD | 18 months

CONTACTS AND LOCATIONS:
Locations (2):
- Nancy University Hospital, Vandœuvre-lès-Nancy, France
- San Raffaele Hospital, Milan, Italy